CLINICAL TRIAL: NCT00556920
Title: A Randomized, Open-label, Single-dose, Three-period, Crossover Study to Demonstrate the Bioequivalence of the Fixed Dose Combination (FDC) of COREG CR™ and Lisinopril to COREG CR and ZESTRIL
Brief Title: Study to Demonstrate the Bioequivalence of the Fixed Dose Combination of COREG CR™ and Lisinopril to Its Components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFD106094
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
Keywords: Coreg CR
MeSH Terms: conditions — Hypertension | interventions — Carvedilol

INTERVENTIONS:
Drug: COREG CR

SUMMARY:
This study will be a randomized study investigating the bioequivalence of COREG CR and Lisinopril to COREG CR and ZESTRIL

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* males and females 18-55 yrs old
* non-orthostatic hypotension
* Body weight > 60 kg (132 lbs) and body mass index (BMI) between 19 and 33 kg/m2

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history, physical or laboratory examination, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Subjects who metabolize carvedilol poorly based on CYP2D6 genotyping as determined at screening.
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements, as well as grapefruit-containing products) within 7 days or 5 half-lives (whichever is longer) prior to first dose of study medication and until the end of the study. Treatment with any CYP2D6 inhibitors such as but not limited to quinidine, fluoxetine, paroxetine, duloxetine, and terbinofine at least 14 days or 5 half-lives (whichever is longer) prior to Day 1 of Session 1 and until the end of the study.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Day 1 of Session 1.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Positive urine drug screen (UDS) including alcohol at screening. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urine Na/creatinine ratio < 0.08 meq/mg.
* Positive for Hepatitis B surface antigen, or HIV.
* Women of child-bearing potential.
* Resting heart rate of ≤ 50 beats per minute (bpm) at screening.
* Abnormalities on 12-lead ECG during screening
* Documented history of low blood pressure (average SBP ≤ 110 mm Hg and/or DBP ≤ 50 mm Hg) or blood pressure below these values at time of screening.
* Orthostatic hypotension diagnosed at screening (orthostatic hypotension will be defined as a reduction in systolic blood pressure of 20 mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing vs. supine measurements. (See Section 6.2.6).
* Donation of blood in excess of 500 mL within a 56-day period including approximately 350 mL of blood to be drawn during this study.
* History of asthma, COPD and/or hypersensitivity to β-adrenergic blocking agents.
* History of sensitivity to heparin, heparin- induced thrombocytopenia, or sensitivity to any of the study medications or components thereof.
* History of anaphylaxis or anaphylactic reactions or severe allergic responses to drugs.
* History of angioedema.
* History of sensitivity to carvedilol, lisinopril, alpha-blockers, beta-blockers or ACE inhibitors.
* Unwillingness or inability to follow the procedures outlined in the protocol or inability to provide written informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood Sampling over a period of 96 hours post dosing of Investigational product in all sessions. Safety: ECG, Vital Signs, clinical labs over 96 hours post dosing. Continuous Adverse event monitoring from dosing until study conclusion and followup. | 96 hours

SECONDARY OUTCOMES:
To assess other pharmacokinetic parameters, evaluate the safety and tolerability Safety: ECG, Vital Signs, Clinical labs over a 96 hour period following dose of investigational product. Continuous adverse event report for ever session | 96 Hours
PK parameters: Tmax and t1/2 of carvedilol [racemate] and lisinopril.
Safety and tolerability will be assessed by clinical data from Adverse Event reporting, nurse/physician observations, vital signs, ECGs, and clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States